CLINICAL TRIAL: NCT05231564
Title: Study of Hybrid Training on Lipid Profile and Non-alcoholic Fatty Liver Disease in Middle-aged Obese Women
Brief Title: Hybrid Training and Middle Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sistan and Baluchestan (Other)
Collaborators: Niloofar Zareie Mohammad Zadeh (Unknown)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, Asst.Prof.Dr. of sports science, University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: no grant
Record Dates: First submitted 2022-01-19; First posted 2022-02-09 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Women's Health; Hybrid Training; Middle Aged; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid training (Experimental): 15 women for hybrid training.
  Interventions: Other: hybrid training
- Healthy lifestyle counseling (No Intervention): 15 women for healthy lifestyle counseling

INTERVENTIONS:
Other: hybrid training — The experimental group trained two to three sessions of 45 to 50 minutes a week with a recovery of 24 to 48 hours between each session to burn 500 kcal. The first three weeks held hybrid training with a metabolic program and the other three weeks held a strength training program.
  Arms: Hybrid training

SUMMARY:
Modern living and physical inactivity results in many ailments, including obesity, non-alcoholic fatty liver disease (NAFLD), and inflammatory issues.

Though there are a lot of studies on physical training, there is little detail on hybrid training or electrical and voluntary contractions of the musculature. This study investigated the efficiency of hybrid training in biochemistry, ultrasound, and proinflammatory outcomes in middle-aged sedentary and obese women with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women with one to two exercise sessions or less per month
* BMI equal to or above 30 kg/m-2
* WHR equal or above 0.85 m
* Confirmed NAFLD, with grade 2 and 3
* Systolic blood pressure not less than 130 mm Hg and diastolic blood pressure not less than 85 mm Hg
* Increased AST and ALT
* Mean age 45-65 years

Exclusion Criteria:

* Use of 140 grams or more of ethanol per week
* History of depression in the last 6 months
* History of chronic or acute viral hepatitis
* Drug-related liver disease and chronic liver disease
* History of diabetes
* Uncontrolled hypertension
* Myocardial infarction
* Chronic kidney disease
* Hyperthyroidism or heart failure
* Those who have weight loss programs or medical contraindications for physical training
* Serious arterial hemorrhagic disorders
* Serious neurological diseases
* Advanced atherosclerosis
* Elevated fever

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The statistical population consisted of sedentary, obese middle-aged women who were not on medication.
Enrollment: 15 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Body Weight | Pre-study
  in kg
Body Mass Index | Pre-study
  in kg/m-2
Aspartate transaminases | Pre-study
  in u/l
Alanine transaminases | Pre-study
  in u/l
Fasting blood sugar | Pre-study
  in mg/dl
Proinflammatory cytokine (interleukin -6) | Pre-study
  in pg/ml
Ultrasonic assessment | Pre-study
  Grade of liver steatosis
WHR | Pre-study
  Waist-to-hip ratio in cm
SBP/DBP | Pre-study
  Systolic blood pressure/Diastolic blood pressure
HDL Cholesterol Plasma | Pre-study
  in mg/dl

SECONDARY OUTCOMES:
Body Weight | six-week
  in kg
Body Mass Index | six-week
  in kg/m-2
Aspartate transaminases | six-week
  in u/l
Alanine transaminases | six-week
  in u/l
Fasting blood sugar | six-week
  in mg/dl
Proinflammatory cytokine (interleukin -6) | six-week
  in pg/ml
Ultrasonic assessment | six-week
  Grade of liver steatosis
WHR | six-week
  Waist-to-hip ratio in cm
SBP/DBP | six-week
  Systolic blood pressure/Diastolic blood pressure
HDL Cholesterol Plasma | six-week
  in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, MD, PhD, Principal Investigator — University of Sistan and Baluchestan
Locations (1):
- Mohammadreza Rezaeipour (MD, PhD), Zahedan, Sistan and Baluchestan, Iran

REFERENCES:
- [Derived] Mohammadzadeh NZ, Rezaeipour M. "Hybrid exercise training improves liver steatosis and inflammation in a randomized trial of sedentary, obese women with non-alcoholic fatty liver disease". BMC Sports Sci Med Rehabil. 2025 Oct 24;17(1):308. doi: 10.1186/s13102-025-01349-2. PMID 41137140